CLINICAL TRIAL: NCT05809154
Title: Prospective Cohort Study of Patients With Lower Urinary Tract Dysfunction Undergoing Urodynamic Examination for the Assessment of Quality, Cost and Treatment Success
Brief Title: Quality, Cost and Treatment Success on Patients With Lower Urinary Tract Dysfunction Undergoing Urodynamic Examination
Acronym: UroLUTS
Status: Withdrawn | Type: Observational
Why Stopped: Personnel changes
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: UroLUTS
Record Dates: First submitted 2018-09-18; First posted 2023-04-12 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Urodynamics; Lower Urinary Tract Symptoms; Neurogenic Bladder
Keywords: Urodynamics; Lower Urinary Tract Symptoms; Neurogenic Bladder
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Bladder, Neurogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Neurogenic lower urinary tract dysfunction: Lower urinary tract dysfunction due to any neurological condition like spinal cord injury, multiple sclerosis and others.
  Interventions: Diagnostic Test: Video-Urodynamics
- Non-Neurogenic lower urinary tract dysfunction: Lower urinary tract dysfunction in absence of any neurological pathology.
  Interventions: Diagnostic Test: Video-Urodynamics
- Chronic pelvic pain: Chronic pelvic pain as defined by the EAU guidelines.
  Interventions: Diagnostic Test: Video-Urodynamics
- Urodynamic normal Bladder function: Normal urodynamic findings and absence of chronic pelvic pain.
  Interventions: Diagnostic Test: Video-Urodynamics

INTERVENTIONS:
Diagnostic Test: Video-Urodynamics — Minimal invasive Urodynamic examination: Cystomanometry for the assessment of the bladder storage phase and a pressure-flow for the assessment of the voiding phase. By a thin transurethral catheter, body warm fluid is filled in to the bladder and at the same time is the intravesical and abdominal pressure traced with a computer system. The pelvic floor muscle activity is assessed at the same time using EMG surface electrodes.

SUMMARY:
Lower urinary tract dysfunction (LUTD) is a very common complication of urological, gynecological, neurological, metabolic, inflammatory or tumor disease. LUTD is not an inevitable condition, the investigators can help in many ways. Modern clinical examinations like urodynamics allow for patient tailored treatment strategies. Urodynamics however, even if minimal invasive, may lead to urinary tract infections and are very expensive4. Aim of this study is to evaluate in the long-term perspective what patients profit of urodynamic examinations and in what patients the investigators could resign to perform urodynamics in the future and or in what patients the interval of urodynamics could be extended. Main objective is to follow in a long-term prospective cohort study, patients suffering of lower urinary tract dysfunction (LUTD). In this observational study the investigators will include all patient undergoing clinical routine urodynamic examination to better address what is the normal course of LUTD with and without Treatment. The aim is to have a prospective urodynamics database allowing to answer questions related to urodynamics.

DETAILED DESCRIPTION:
Patients with a clinical indication for routine urodynamic assessment will be included in to this prospective cohort study. All standard urodynamic results as well as the treatment decision will be collected. Patients undergoing repeated urodynamic measurements i.e. spinal cord injured patients with yearly assessments will each time be included allowing for long-term and follow up analysis of both disease progress and therapy success.

Bladder function is rather simple: storage and voiding of urine. The control of the urinary bladder on the other hand is very complex with many areas that still remain unclear, as for example the cross play of the central and and autonomous nervous system. Voiding of the bladder is an active process that is controlled by nervous impulses from the central nervous system. The detrusor muscle is contracted, and the urethral sphincter muscle is relaxed at the same time so that the urine can be drained off.

Uroflow examination in combination with post-void residual assessment (by sonography or catheterization) are a simple but powerful screening tool to evaluate bladder function. Since both the uroflow as well as the post-void residual are dependent on the detrusor pressure and the infravesical resistance they do not allow for differentiation between hypocontractile detrusor muscle and infravesical obstruction or a combination of both. To do so, the minimal invasive Urodynamic examination is needed. Cystomanometry for the assessment of the bladder storage phase and a pressure-flow for the assessment of the voiding phase. By a thin transurethral catheter, body warm fluid is filled in to the bladder and at the same time is the intravesical and abdominal pressure traced with a computer system. The pelvic floor muscle activity (i.e. the urethral sphincter muscle) is assessed at the same time using EMG surface electrodes.

For Video-Urodynamics, Contrast agent is mixed in to the body warm infusion solution allowing to judge bladder configuration (i.e. diverticula or trabeculation) and if there is vesico-uretero-renal reflux.

Patients with a clinical indication for routine urodynamic assessment will be included in to this prospective cohort study. All standard urodynamic results as well as the treatment decision will be collected. Patients undergoing repeated urodynamic measurements i.e. spinal cord injured patients with yearly assessments will each time be included allowing for long-term and follow up analysis of both disease progress and therapy success.

Except for urinary tract infections, are complications in urodynamic measurements very rare. The investigators estimate additional complications (like pain or autonomic dysreflexia) in about 1% of urodynamic examinations. To have a minimum of 50 complications, the investigators aim to include about 5000 urodynamic examinations for reliable numbers of each complication, ideally allowing for subgroup analysis.

All patients undergoing clinical routine urodynamic examination will be included, i.e. per year approximately 500 urodynamic measurements and 450 patients (some patients will have multiple measurements per year). With the aim of 5000 included urodynamic examinations the investigators estimate a study duration of 10 years. This has the advantage that the investigators will also have a meaningful average follow-up of at least 5 years or more in patients undergoing annual urodynamic measurements (e.g. spinal cord injured patients).

Descriptive statistics: Data will be presented on interval-scales with median and quartiles or with means and standard deviations summarized. Dichotomic variables will be presented as ratios and percentages.

Univariate analysis: t-test will be used to compare means between groups and Chi-Square for the comparison of dichotomic variables.

Multivariate analysis: To assess the distribution of initial parameters the investigators will use multivariate regression models.

ELIGIBILITY:
Inclusion Criteria:

* Participants fulfilling all of the following inclusion criteria are eligible for the study:

  * Female and male patients, age >18 years
  * Informed consent
  * Lower urinary tract symptoms
  * Planned clinical routine urodynamic examination

Exclusion Criteria:

* The presence of any of the following exclusion criteria will lead to exclusion of the participant:

  * Age <18 years
  * Pregnancy or breast feeding
  * Individuals especially in need of protection (according to Research with Human Subjects published by the Swiss Academy of Medical Sciences https://www.samw.ch/en/Publications/Medical-ethical-Guidelines.html)
  * No informed consent
  * Patients incapable to follow the trial, e.g. because of language problems, psychiatric disorders, dementia and so on.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a clinical indication for routine urodynamic assessment will be included in to this prospective cohort study. All standard urodynamic results as well as the treatment decision will be collected. Patients undergoing repeated urodynamic measurements i.e. spinal cord injured patients with yearly assessments will each time be included allowing for long-term and follow up analysis of both disease progress and therapy success.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Number of voids per 24 hours | At the urodynamic assessment, up to 24 hours
  Number of voids per 24 hours
Number of leakages per 24 hours | At the urodynamic assessment, up to 24 hours
  Number of leakages per 24 hours
Number of used pads per 24 hours | At the urodynamic assessment, up to 24 hours
  Number of used pads per 24 hours
Post void residual (mL) | At the urodynamic assessment, up to 10-30 minutes
  Residual urine remaining in the bladder after voiding.

SECONDARY OUTCOMES:
Cystometric capacity (mL) | At the urodynamic assessment, up to 10-30 minutes
  Measured in mL in urodynamics
Compliance (mL/cmH2O) | At the urodynamic assessment, up to 10-30 minutes
  Measured in mL/cmH2O in urodynamics
Bladder volume (mL) at detrusor overactivity | At the urodynamic assessment, up to 10-30 minutes
  Measured in mL in urodynamics
Maximum detrusor pressure amplitude (cmH2O) at detrusor overactivity | At the urodynamic assessment, up to 10-30 minutes
  Measured in cmH2O in urodynamics
Detrusor leak point pressure (cmH2O) | At the urodynamic assessment, up to 10-30 minutes
  Measured in cmH2O in urodynamics
Maximum detrusor pressure (cmH2O) during storage phase | At the urodynamic assessment, up to 10-30 minutes
  Measured in cmH2O in urodynamics
Maximum detrusor pressure (cmH2O) during voiding phase | At the urodynamic assessment, up to 10-30 minutes
  Measured in cmH2O in urodynamics
Detrusor pressure at maximum flow | At the urodynamic assessment, up to 10-30 minutes
  Measured in urodynamics
Scores in Qualiveen & International Prostate Symptom Score (IPSS) | At the urodynamic assessment, up to 10-30 minutes
  Score value between 0 and a maximum of 35 points. Interpretation: Mild (IPSS<8), moderate (IPSS=8-19) and severe (IPSS=20-35) symptoms
Scores in Female Sexual Function Index (FSFI) | At the urodynamic assessment, up to 10-30 minutes
  The FSFI1 is a 19-item, self-report measure of female sexual function that provides scores on overall levels of sexual function as well as the primary components of sexual function in women, including sexual desire, arousal, orgasm, pain, and satisfaction. To score the measure of 19 Items, the sum of each domain score is first multiplied by a domain factor ratio (0.6 for desire; 0.3 for arousal; 0.3 for lubrication; 0.4 for orgasm; 0.4 for satisfaction; and 0.4 for pain) in order to place all domain totals on a more comparable scale, and then subsequently summed to derive a total FSFI score. The absence of sexual activity or intercourse is not necessarily attributable to sexual dysfunction. proper scoring and interpretation of the measure necessitates: a) inclusion of a distress measure for diagnosing sexual dysfunction clinically, as defined by current standards; and b) correction for sexual activity status and adapted scoring for sexually inactive respondents.
Number of patients with adverse events grade 1 bis 5 following the National Cancer Institute terminology Vers. 4 (Common Terminology Criteria for Adverse Events (CTCAE) | At the urodynamic assessment, up to 10-30 minutes
  urodynamic assessment
International Index of Erectile Function (IIEF) | At the urodynamic assessment, up to 10-30 minutes
  Based on IIEF, ED severity is classified into five categories: no ED (score 22-25), mild (17-21), mild to moderate (12-16), moderate (8-11), and severe (5-7).

CONTACTS AND LOCATIONS:
Overall Officials: Marc P Schneider, MD, PhD, Study Chair — Universitätsklinik für Urologie

IPD SHARING:
Plan to Share IPD: No
We do not share IPD with other researchers.